CLINICAL TRIAL: NCT03824171
Title: A Randomized, Open Label, Single Dose, Crossover Study to Evaluate the Safety and Pharmacokinetic Characteristics After Administration of AD-102 in Healthy Male Subjects
Brief Title: Evaluating the Pharmacokinetic Characteristics of AD-102 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AD-102BE
Record Dates: First submitted 2019-01-28; First posted 2019-01-31 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Raloxifene Hydrochloride; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Raloxifene 60mg/Cholecalciferol 800IU to AD-102 (Experimental): Period 1: Raloxifene 60mg/Cholecalciferol 800IU, 2 tab, QD, Per oral Period 2: Raloxifene 45mg/Cholecalciferol 800IU, 2 tab, QD, Per oral
  Interventions: Drug: Raloxifene 60mg/Cholecalciferol 800IU; Drug: AD-102
- AD-102 to Raloxifene 60mg/Cholecalciferol 800IU (Experimental): Period 1: Raloxifene 45mg/Cholecalciferol 800IU, 2 tab, QD, Per oral Period 2: Raloxifene 60mg/Cholecalciferol 800IU, 2 tab, QD, Per oral
  Interventions: Drug: Raloxifene 60mg/Cholecalciferol 800IU; Drug: AD-102

INTERVENTIONS:
Drug: Raloxifene 60mg/Cholecalciferol 800IU — Raloxifene 60mg/Cholecalciferol 800IU tablet
Drug: AD-102 — AD-102 Raloxefene 45mg/Cholecalciferol 800IU tablet

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic characteristics of AD-102 in healthy male subjects

DETAILED DESCRIPTION:
This study is to evaluate the pharmacokinetic characteristics and safety of AD-102 compared with administration of raloxifen 60 mg + Cholecalciferol 800IU in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 17.5 kg/m2 and 30.5 kg/m2 at the time of screening visit
* The Age between 19 and 50 in healthy male volunteers at the time of screening visit

Exclusion Criteria:

* As a result of laboratory tests, the following figures: ALT or AST> 2 times upper limit of normal range
* As a result of laboratory tests, the following figures: 25-OH vitamin D total <9 ng/mL

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | pre-dose to 96 hours
  Cmax of Raloxifene
Peak Plasma Concentration (Cmax) | pre-dose to 72 hours
  Cmax of corrected Cholecalciferol
Area under the curve in time plot (AUCt) | pre-dose to 96 hours
  AUCt of Raloxifene
Area under the curve in time plot (AUCt) | pre-dose to 72 hours
  AUCt of corrected Cholecalciferol

SECONDARY OUTCOMES:
Area under the curve in time plot (AUCinf) | pre-dose to 96 hours
  AUCinf of Raloxifene
Area under the curve in time plot (AUCinf) | pre-dose to 72 hours
  AUCinf of Corrected Cholecalciferol
Time to reach Cmax | pre-dose to 96 hours
  Tmax of Raloxifene
Time to reach Cmax | pre-dose to 72 hours
  Tmax of Corrected Cholecalciferol
Effective half-life | pre-dose to 96 hours
  t1/2 of Raloxifene
Effective half-life | pre-dose to 72 hours
  t1/2 of Corrected Cholecalciferol

OTHER OUTCOMES:
Number of participants with adverse events | From Day 1 until 32 Days
  Incidence rate of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hosptial, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No